CLINICAL TRIAL: NCT06173076
Title: A Prospective Study to Evaluate Clinical Outcomes in Patients With Anti-leucine-rich Glioma-inactivated 1 Encephalitis
Brief Title: A Prospective Study to Evaluate Clinical Outcomes in Anti-LGI1 Encephalitis
Status: Recruiting | Type: Observational
Sponsor: Shen Chun-Hong (Other)
Responsible Party: Sponsor-Investigator, Shen Chun-Hong, Associate Senior Doctor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Other Study IDs: Y2022-0336
Record Dates: First submitted 2023-11-14; First posted 2023-12-15 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Encephalitis; Leucine-Rich Glioma Inactivated 1 Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and cerebrospinal fluid samples will be stored to test antibodies, cytokines, immune cells and other relevant molecules. And patients have the right to destroy them at any time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Anti-leucine-rich glioma-inactivated 1 (LGI1) encephalitis has been increasingly identified as the second most common type of autoimmune encephalitis after anti-N-methyl-D-aspartate receptor (NMDAR) encephalitis. It presents with acute or subacute onset of epileptic seizures, anterograde amnesia, behavior disturbances, sleep disorders and hyponatremia. In most patients with anti-LGI1 encephalitis, immunotherapy is successful in treating the encephalitis. However, relapses, chronic epilepsy, cognitive declines and psychiatric problems have been reported in some cases.

So far, prospective studies to evaluate its clinical outcomes still remain limited. In this project, the investigators will use clinical features and advanced paraclinical examinations to prospectively investigate the clinical outcomes and the associated factors in patients with anti-LGI1 encephalitis.

DETAILED DESCRIPTION:
In this prospective study, the investigators are aiming to recruit newly diagnosed patients with anti-LGI1 encephalitis. At the acute stage and during the follow-up, some routine and advanced paraclinical examinations will be conducted, including dynamic blood and/or cerebrospinal fluid (CSF) test, multimodal brain magnetic resonance imaging (MRI) including functional MRI, diffusion tensor imaging, arterial spin labeling, et al), Electroencephalography (EEG) or continuous video-EEG (VEEG), positron emission tomography (PET), neuropsychological tests and some other paraclinical examinations. Through the comprehensive analysis, the clinical outcomes and associated factors are further explored in anti-LGI1 encephalitis.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the 2016 consensus diagnostic criteria for anti-LGI1 encephalitis.
2. Newly diagnosed, and during the acute stage before study enrollment.
3. Sign the informed consent form.

Exclusion Criteria:

1. with the diagnosis of epilepsy, stroke, cerebral trauma, and/or other nervous system disease prior to the onset of encephalitis.
2. with coexisting antibodies, such as anti-contactin-associated protein 2 (CASPR2) antibody.
3. Lost to follow-up.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients with anti-LGI1 encephalitis
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
seizure outcomes | 1 year, 2 year
  The incidence of different seizure outcomes and associated factors will be analyzed.
Clinical severity and recovery 1 | 1 year, 2 year
  modified Rankin scale, ranging from 0-6, higher scores mean a worse outcome
Clinical severity and recovery 2 | 1 year, 2 year
  clinical assessment scale for autoimmune encephalitis, ranging from 0-27, higher scores mean a worse outcome
Incidence of recurrence | 1 year, 2 year
  a relapse of encephalitis

SECONDARY OUTCOMES:
Memory assessment 1 | 1 year, 2 year
  the Wechsler Memory Scale, high score means a good memory.
Memory assessment 2 | 1 year, 2 year
  Rey Auditory Verbal Learning Test (RAVLT), high score means a good vebal episodic memory.
Brain volume | 1 year, 2 year
  with 3T magnetic resonance imaging (MRI), volumes of the whole hippocampus, hippocampal subfields and other relevant regions were determined using FreeSurfer. The unit of volume is described as mm3.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hong Shen, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No